CLINICAL TRIAL: NCT05574608
Title: Early Clinical Study of Allogenic CD123-CAR-NK Cells (JD023 Injection) in the Treatment of Refractory or Relapsed CD123-positive Acute Myeloid Leukemia
Brief Title: Allogenic CD123-CAR-NK Cells in the Treatment of Refractory/Relapsed Acute Myeloid Leukemia
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Affiliated Hospital to Academy of Military Medical Sciences (Other)
Collaborators: Beijing JD Biotech Co. LTD. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CAR-NK123-JD
Record Dates: First submitted 2022-09-28; First posted 2022-10-10 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Acute Myeloid Leukemia Refractory; Acute Myeloid Leukemia Recurrent

STUDY DESIGN:
Intervention Model Description: Evaluate the safety of JD023 injection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Experimental: CD123-CAR-NK. (Experimental): The relapsed/refractory AML patients will receive allogenic CD123-Targeted CAR-NK cells infusion (1x10^9, 1-2x10^7/kg) after precondition chemotherapy.
  Interventions: Biological: CD123-CAR-NK cells

INTERVENTIONS:
Biological: CD123-CAR-NK cells — CD123-CAR-NK is an allogenic CD123-Targeted chimeric antigen receptor NK-cell (CAR-NK) therapy.

SUMMARY:
The CD123-Targeted CAR-NK cell therapy is a new treatment that is being investigated for treatment of acute myeloid leukemia (AML). The purpose of this study is to evaluate the safety of CD123-CAR NK cells given to these patients.

DETAILED DESCRIPTION:
This is a study of allogenic CD123-CAR NK cells. The relapsed/refractory AML patients will receive FC (F, Fludarabine, C, Cyclophosphamide) chemotherapy followed by infusion of CD123-CAR-NK cells. No graft-versus-host disease (GVHD) prevention will be conducted before or after infusion. Dose-limiting toxicity, incidence of adverse events, disease response and PK/PD will be detected post-infusion.

ELIGIBILITY:
Inclusion criteria:

1. Age ≥ 18 years old, no gender or race;
2. Expected survival period ≥ 3 months;
3. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 2;
4. The diagnosis of AML with bone marrow biopsy, immunohistochemistry or Flow cytometry definitively positive for CD123 and met one of the following criteria:

   A. Diagnostic criteria for relapsed AML: after complete remission (CR), leukemia cells reappeared in peripheral blood or blast cells in bone marrow ≥ 5% (except for other reasons such as bone marrow regeneration after consolidation chemotherapy) or extramedullary leukemia cell infiltration; B. Diagnostic criteria for refractory AML: naive patients who were ineffective after 2 courses of standard regimens; patients relapsed within 12 months who underwent consolidation and intensive therapy after CR; patients relapsed after 12 months but were ineffective after conventional chemotherapy; Patients with two or more relapses; patients with persistent extramedullary leukemia; C. Patients eligible for relapsed or refractory AML remained minimally residual disease positive after salvage therapy
5. Adequate organ function:

   A. Liver function: ALT≤3×ULN, AST≤3×ULN, total bilirubin≤2×ULN; B. Coagulation function: international normalized ratio (INR) or activated partial thromboplastin time (APTT) ≤ 1.5×ULN; C. Renal function: serum creatinine≤1.5×ULN or creatinine clearance rate ≥30mL/min; D. Cardiac function: Left ventricular ejection fraction (LVEF) ≥ 50%;
6. Women of child-bearing potential and all male participants must use effective methods of contraception for at least 12 months after infusion.;
7. Informed Consent/Assent: All subjects must have the ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

1. Central nervous system involved;
2. Known contraindication to the protocol defined lymphodepleting chemotherapy regimen of fludarabine/cyclophosphamide;
3. Systemic use of hormones within 2 weeks prior to enrollment (except for patients with inhaled corticosteroids);
4. Any active infection requiring systemic therapy by intravenous infusion within 14 days prior to the first dose of study drug, including: HBV, HCV, HIV, syphilis infection, or active pulmonary tuberculosis.
5. History of hypersensitivity reactions to murine protein-containing products, or macromolecular biopharmaceuticals such as antibodies or cytokines;
6. Patients cannot guarantee effective contraception (condom or contraceptives, etc.) within 1 years after enrollment;
7. Women who are pregnant (urine/blood pregnancy test positive) or lactating;
8. Suffering from a serious autoimmune disease or immunodeficiency disease; 9 Suffering from mental illness;

10. Known alcohol dependence or drug dependence; 11. According to the investigator's judgment, the patient has other unsuitable grouping conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicities (DLTs) | 1 Months
Treatment-emergent adverse events | 3 months
Treatment-related adverse events | 3 months

SECONDARY OUTCOMES:
Complete response (CR) | 3 months
Progression free survival (PFS) | 12 months
Overall Survival (OS) | 12 months
Proportion of subjects with minimal-residual disease (MRD) negative response | 3 months
The area under the concentration time-curve (AUC) of CD123-CAR-NK cells | 3 Months
Peak levels of CD123-CAR-NK cells (maximum concentration or Cmax) | 3 Months

CONTACTS AND LOCATIONS:
Overall Officials: Liangding Hu, Docotr, Principal Investigator — The Fifth Medical Center of Chinese People's Liberation Army (PLA) General Hospital, Beijing, China.
Locations (1):
- The Fifth Medical Center of Chinese People's Liberation Army (PLA) General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No